CLINICAL TRIAL: NCT03004248
Title: An Open-Label, Multi-Center Trial to Assess the Safety of Single and Repeat Treatments of DaxibotulinumtoxinA for Injection for Treatment of Moderate to Severe Glabellar Lines (SAKURA OPEN-LABEL SAFETY)
Brief Title: Safety of Single and Repeat Treatments of DaxibotulinumtoxinA for Injection for Treatment of Moderate to Severe Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1620303
Record Dates: First submitted 2016-12-22; First posted 2016-12-28 (Estimated); Results first posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-06

CONDITIONS: Glabellar Frown Lines
Keywords: glabellar lines, frown lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DaxibotulinumtoxinA 40 units (Experimental): Biological/Vaccine: Botulinum Toxins, Type A Intramuscular injection
  Interventions: Biological: Botulinum Toxins, Type A

INTERVENTIONS:
Biological: Botulinum Toxins, Type A — Intramuscular Injection
  Other Names: DaxibotulinumtoxinA

SUMMARY:
This is a long term safety study of DaxibotulinumtoxinA for Injection for the treatment of moderate to severe glabellar lines following single and repeat administration.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent including authorization to release health information
* Moderate (2) or severe (3) glabellar lines during maximum frown based on the Investigator Global Assessment Frown Wrinkle Severity (IGA-FWS) scale
* Moderate (2) or severe (3) glabellar lines during maximum frown based on the Patient Frown Wrinkle Severity (PFWS) scale
* Willing and able to follow all trial procedures, attend all scheduled visits, and successfully complete the trial

Exclusion Criteria:

* Any neurological condition that may place the subject at increased risk with exposure to botulinum toxin type A, including peripheral motor neuropathic diseases such as amyotrophic lateral sclerosis and motor neuropathy, and neuromuscular junctional disorders such as Lambert-Eaton syndrome and myasthenia gravis
* Active skin disease, infections or inflammation at the injection sites
* Plan to receive botulinum toxin type A anywhere in the face through the duration of the study
* History of allergy or sensitivity to any botulinum toxin preparations or to any component of the test article
* Current enrollment in an investigational drug or device trial or participation in such a trial within the last 30 days prior to screening through end of trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2691 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (52):
- United States (47):
  - Birmingham, Alabama
  - Beverly Hills, California
  - Encinitas, California
  - Fremont, California
  - Los Angeles, California
  - Manhattan Beach, California
  - Newport Beach, California
  - Roseville, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Santa Monica, California
  - Greenwood Village, Colorado
  - Washington D.C., District of Columbia
  - Boca Raton, Florida
  - Bradenton, Florida
  - Coral Gables, Florida
  - Miami, Florida
  - West Palm Beach, Florida
  - Chicago, Illinois
  - Lincolnshire, Illinois
  - Naperville, Illinois
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Glenn Dale, Maryland
  - Hunt Valley, Maryland
  - Rockville, Maryland
  - Chestnut Hill, Massachusetts
  - Birmingham, Michigan
  - Fridley, Minnesota
  - St Louis, Missouri
  - Omaha, Nebraska
  - Montclair, New Jersey
  - New York, New York
  - West Islip, New York
  - White Plains, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - High Point, North Carolina
  - Portland, Oregon
  - Drexel Hill, Pennsylvania
  - Nashville, Tennessee
  - Austin, Texas
  - College Station, Texas
  - Houston, Texas
  - Katy, Texas
  - Mequon, Wisconsin
- Canada (5):
  - Vancouver, British Columbia
  - Burlington, Ontario
  - Toronto, Ontario
  - Woodbridge, Ontario
  - Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Green JB, Mariwalla K, Coleman K, Ablon G, Weinkle SH, Gallagher CJ, Vitarella D, Rubio RG. A Large, Open-Label, Phase 3 Safety Study of DaxibotulinumtoxinA for Injection in Glabellar Lines: A Focus on Safety From the SAKURA 3 Study. Dermatol Surg. 2021 Jan 1;47(1):42-46. doi: 10.1097/DSS.0000000000002463. PMID 32773447
- [Derived] Fabi SG, Cohen JL, Green LJ, Dhawan S, Kontis TC, Baumann L, Gross TM, Gallagher CJ, Brown J, Rubio RG. DaxibotulinumtoxinA for Injection for the Treatment of Glabellar Lines: Efficacy Results From SAKURA 3, a Large, Open-Label, Phase 3 Safety Study. Dermatol Surg. 2021 Jan 1;47(1):48-54. doi: 10.1097/DSS.0000000000002531. PMID 32773446

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Outpatient, male or non-pregnant, non-nursing females, 18 years of age or older, and in good general health with moderate (2) or severe (3) glabellar lines during maximum frown based on the IGA-FWS and PFWS.
Period: Overall Study
Arm/Group | DaxibotulinumtoxinA 40 Units
Started | 2691
Received a Single Treatment | 1809
Received Two Treatments | 314
Received Three Treatments | 568
Completed | 2314
Not Completed | 377

BASELINE CHARACTERISTICS:
Population: Safety population consisting of all enrolled subjects.
Arm/Group | DaxibotulinumtoxinA 40 Units
Number analyzed (Participants) | 2691
Age, Continuous [Median (Full Range); unit: years] | 50.0 [21 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2383
  Male | 308
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 2407
  Race: Black of African American | 129
  Race: Others | 82
  Race: Asian | 73
Region of Enrollment [Number; unit: participants]
  North America | 2691

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment Emergent Adverse Events (TEAE)
Description: Incidence rates based on the number and percentage of subjects treated within each cycle who report Adverse Events (AEs) at anytime following study treatment. Note that subjects could receive up to 3 consecutive treatments during the 36-week follow up period.
Time Frame: 0-36 weeks
Population: Safety Evaluable Population
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Cycle 1; Treatment Cycle 2; Treatment Cycle 3: Biological/Vaccine: Botulinum Toxins, Type A Intramuscular injection
  Botulinum Toxins, Type A: Intramuscular Injection
Arm/Group | Treatment Cycle 1 | Treatment Cycle 2 | Treatment Cycle 3
Number analyzed (Participants) | 2380 | 882 | 568
Participants | 831 | 267 | 118

2. Secondary Outcome: Percentage of Subjects Who Achieved ≥ 2 Point Improvement Independently and Concurrently on Investigator and Patient Rating Scales
Description: Percentage of subjects who achieve at least a 2-point improvement from baseline and a score of 0 or 1 (i.e. none or mild wrinkles in severity) on both Investigator and Subject Frown Wrinkle Severity (FWS) assessments
Time Frame: Week 4
Population: Safety Evaluable Population
Measure: Number; unit: percentage of responders
Arm/Group | Treatment Cycle 1 | Treatment Cycle 2 | Treatment Cycle 3
Number analyzed (Participants) | 2380 | 882 | 568
percentage of responders | 73.2 | 76.8 | 76.6

3. Secondary Outcome: The Time to Return to Moderate to Severe on Both IGA-FWS and PFWS Scales for DaxibotulinumtoxinA for Injection Group
Description: The time to return to moderate to severe on both scales was measured following treatment cycles 1 and 2. Because subjects were only followed for 12 weeks following treatment cycle 3, time to return was not analyzed for this cycle.
Time Frame: 0-36 weeks per cycles 1 and 2
Population: Safety Evaluable Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment Cycle 1 | Treatment Cycle 2
Number analyzed (Participants) | 2380 | 882
days | 168.0 [167 to 168] | 169.0 [168 to 173]

4. Secondary Outcome: The Time to Return to, or Worse Than, Baseline on Both IGA-FWS and PFWS Scales for DaxibotulinumtoxinA for Injection Group
Description: The time to return to or worse than baseline on both FWS scales was measured following treatment cycles 1 and 2. Because subjects were only followed for 12 weeks following treatment cycle 3, time to return was not analyzed in this cycle.
Time Frame: 0-36 weeks per Cycle 1 and 2
Population: Safety Evaluable Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment Cycle 1 | Treatment Cycle 2
Number analyzed (Participants) | 2380 | 882
days | 196 [196 to 197] | 197 [196 to 199]

ADVERSE EVENTS:
Time Frame: 0-54 weeks
Description: Does not differ than the Clinicaltrials.gov definition
Groups:
- Overall: Biological/Vaccine: Botulinum Toxins, Type A Intramuscular injection
  Botulinum Toxins, Type A: Intramuscular Injection
Arm/Group | Overall
All-Cause Mortality (participants affected / at risk) | 1/2691
Serious Adverse Events (participants affected / at risk) | 29/2691
Other Adverse Events (participants affected / at risk) | 158/2691
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=2691)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Pancreatis acute (Gastrointestinal disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Invasive ductal breat carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Optic neuritis (Nervous system disorders) | 1 (1)
Parasthesia (Nervous system disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Adenomyosis (Reproductive system and breast disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=2691)
Headache (Nervous system disorders) | 158 (183)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
With respect to any proposed publication or disclosure of the results of the Study, the Study Center and Investigator shall submit to Revance a copy of the proposed publication or disclosure at least sixty (60) days prior to the submission thereof for publication or disclosure to a third party: (i) to provide Revance with the opportunity to review and comment on the contents thereof, and (ii) to identify any Confidential Information to be deleted from the proposed publication or disclosure.

DOCUMENTS (2):
  • Study Protocol (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT03004248/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT03004248/SAP_001.pdf